CLINICAL TRIAL: NCT00404027
Title: Patient and Provider Attitudes in the Healthcare Context
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IIR 04-201
Record Dates: First submitted 2006-11-22; First posted 2006-11-27 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to assess patient and provider attitudes towards the role that patients should play in medical decision making and self-management. We will examine the degree to which similarity of attitudes held by VA patients being treated for co-morbid diabetes mellitus and hypertension and by their primary care providers is a determinant of patient satisfaction, patient adherence, and adequacy of blood pressure and diabetic control.

DETAILED DESCRIPTION:
Previous work has shown that similarities in patients' and providers' beliefs about the role each should play in health care contexts are associated with greater patient satisfaction, greater trust in the provider, and greater treatment adherence. Extending this work by examining the effect of patient-provider attitudinal similarity on patients' diabetic and blood pressure control over an 18 month period is important because management of patients with co-morbid hypertension (HTN) and diabetes (DM) is a costly and clinically challenging task within the VA health system. Self-report questionnaires will be used to assess VA providers' beliefs about their own preferences for patient-provider role orientation in care, whereas interviews will be used to measure veterans' beliefs about their preferences for patient-provider role orientation in their care, satisfaction with their care, and self-reported treatment adherence. Data regarding health services use, prescription refills (a measure of adherence), and 18-month means of blood pressure and hemoglobin A1c will be collected from veterans' medical records. The study represents a critical step toward understanding how patient and provider attitudes toward care might be explicitly assessed and incorporated into the evidence-based health care delivery process to enhance the management of chronic illnesses and overall health among veterans.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled in primary care clinics at the study sites (Iowa City VAMC, Jesse Brown VAMC - Chicago) who are scheduled to be seen by a participating provider in the next three (3) months and have been seen on at least three (3) additional occasions by that same

provider in the prior 24 months. Participating patients must also:

i) have prior diagnoses of both HTN and DM, as documented in VA administrative files;

ii) have an active prescription for an anti-hypertensive medication in the following medication classes: thiazide diuretic, beta blocker, angiotensin converting enzyme (ACE) inhibitor, angiotensin receptor blocker (ARB), calcium channel blocker, or alpha blocker;

iii) have an active prescription for an oral hypoglycemic agent or for an insulin preparation;

iv) be able to provide informed consent;

v) have a home telephone; and

vi) reside in an independent living environment and not in a skilled care facility.

Exclusion Criteria:

i) cognitive impairment;

ii) severe underlying illness, including: metastatic cancer, active treatment for any malignancy (excluding basal and squamous cell skin cancers), end-stage renal disease, cirrhosis, severe chronic obstructive lung disease requiring home oxygen therapy, and congestive

heart failure with a documented left ventricular ejection fraction of less than 35% or a prior echocardiogram denoting "severe" left ventricular dysfunction; and

iii) visits in the prior 18 months to a VA endocrinology, cardiology, or nephrology clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veteran primary care patients
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2007-06-04 (Actual); Primary Completion 2010-10-01 (Actual); Study Completion 2010-10-01 (Actual)

PRIMARY OUTCOMES:
PPOS scores | same day as appointment with provider
  Patient-Practitioner Orientation Scale: degree of symmetry between patient and provider regarding patient-centeredness

SECONDARY OUTCOMES:
Blood pressure | Same day as appointment with provider
  Blood pressure measured at time of provider visit
Hemoglobin A1c | Same day as appointment with provider
  Hemoglobin A1c, to assess glycemic control

CONTACTS AND LOCATIONS:
Overall Officials: Alan J. Christensen, PhD, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (1):
- Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa, United States

REFERENCES:
- [Result] Baldwin AS, Vander Weg MW, Christensen AJ, Rothman AJ. Examining the Causal Mechanisms Underlying Self-generated Arguments for Health Behavior Change. [Abstract]. Annals of behavioral medicine : a publication of the Society of Behavioral Medicine. 2009 Apr 1; 37(S):229.
- [Result] Cvengros JA, Christensen AJ, Hillis SL, Rosenthal GE. Patient and physician attitudes in the health care context: attitudinal symmetry predicts patient satisfaction and adherence. Ann Behav Med. 2007 Jun;33(3):262-8. doi: 10.1007/BF02879908. PMID 17600453
- [Result] Baldwin AS, Cvengros JA, Christensen AJ, Ishani A, Kaboli PJ. Preferences for a patient-centered role orientation: association with patient-information-seeking behavior and clinical markers of health. Ann Behav Med. 2008 Feb;35(1):80-6. doi: 10.1007/s12160-007-9011-x. PMID 18347907
- [Result] Cvengros JA, Christensen AJ, Cunningham C, Hillis SL, Kaboli PJ. Patient preference for and reports of provider behavior: impact of symmetry on patient outcomes. Health Psychol. 2009 Nov;28(6):660-7. doi: 10.1037/a0016087. PMID 19916633
- [Result] Howren MB, Christensen AJ, Karnell LH, Funk GF. Health-related quality of life in head and neck cancer survivors: impact of pretreatment depressive symptoms. Health Psychol. 2010 Jan;29(1):65-71. doi: 10.1037/a0017788. PMID 20063937
- [Result] Christensen AJ, Howren MB, Hillis SL, Kaboli P, Carter BL, Cvengros JA, Wallston KA, Rosenthal GE. Patient and physician beliefs about control over health: association of symmetrical beliefs with medication regimen adherence. J Gen Intern Med. 2010 May;25(5):397-402. doi: 10.1007/s11606-010-1249-5. Epub 2010 Feb 20. PMID 20174972